CLINICAL TRIAL: NCT03155035
Title: Effect of Routine Deworming on Weight of Children 5-16 Years Old in an Urban Slum of Karachi: a Randomized Controlled Trial
Brief Title: Effect of Routine Deworming on Weight of Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dow University of Health Sciences (Other)
Responsible Party: Principal Investigator, Zainab Hasan, Principal Investigator, Dow University of Health Sciences
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: IRB-816/DUHS/Approval/2016/351
Record Dates: First submitted 2017-05-14; First posted 2017-05-16 (Actual); Last update posted 2017-07-13 (Actual); Status verified 2017-07

CONDITIONS: Soil Transmitted Helminths
Keywords: deworming; STH
MeSH Terms: interventions — Albendazole; Calcium; Vitamin D

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Albendazole 200 mg 2 tablets single dose
  Interventions: Drug: Albendazole
- Placebo (Placebo Comparator): Calcium 400 mg + vitamin D 2.5 mcg 2 tablets single dose
  Interventions: Dietary Supplement: Calcium 400 mg + Vitamin D 2.5 mcg

INTERVENTIONS:
Drug: Albendazole — Albendazole 400 mg chewable tablets (200 mg each) Two tablets as a single dose recommended as ovicidal, larvicidal and vermicidal against all soil transmitted helminths
  Arms: Intervention
Dietary Supplement: Calcium 400 mg + Vitamin D 2.5 mcg — 2 chewable tablets provide recommended daily allowance for calcium and vitamin D
  Arms: Placebo

SUMMARY:
Soil Transmitted Helminths (STH) are among the most common infections in the world today. The World Health Organization (WHO) recommends mass administration of deworming medicine as a single routine annual dose to all school age children (SAC)(age 5-16 years) in countries where prevalence of Soil Transmitted Helminthic Infections (STHI) is > 20% as a safe public health intervention that promotes healthy growth (Category 2 Recommendation). Pakistan is classified as a low burden community with a reported prevalence of STHI <50%, however,routine deworming is not a policy in Pakistan. Currently, Pakistan is also facing a huge burden of malnutrition in all age groups especially in population belonging to low socioeconomic group. Incidentally, worm infestation by STH also occurs in this group due to associated lack of hygiene and poor living conditions. The coexistence of even moderate STH infections can cause or aggravate malnutrition. The urban slums of Karachi provide environmental, social and behavioral conditions that favor both STH infections and a risk of under nutrition. It is unknown if administering routine dose of deworming medicine to SAC as per WHO recommendation will contribute to improvement in indicators of nutrition status in Pakistani children living in urban slum conditions by eliminating worm infection.Therefore, this study is being conducted to determine the effect of deworming on weight of School Age Children aged between 5 to 16 years.

DETAILED DESCRIPTION:
A randomized control trial will be conducted in an urban slum of Karachi. Eligible 5 to 16 year old school age children will be enrolled after parental consent. The calculated total sample size is n= 258. Subjects will be visited at home by researcher and background information, risk factor presence and baseline measurements of weight, Mid Upper Arm Circumference (MUAC) and tricep skinfold thickness (TSF) will be measured. The intervention arm will be administered a single dose of chewable Albendazole 400 mg and the placebo arm will receive 400 mg chewable calcium tablets. The weight, MUAC and TSF will be measured again after 8 weeks to determine the change if any. The selection of locality and allocation of intervention will be done using simple random sampling and computer generated random numbers.

ELIGIBILITY:
Inclusion Criteria:

* Aged 5 - 16 years, Healthy, Able to chew/swallow tablets

Exclusion Criteria:

* Acutely ill
* Previous deworming dose < 6 months ago
* Intellectually challenged or physical condition interfering with measurement of primary outcome variables

Ages: 5 Years to 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 300 (Actual)
Dates: Start 2017-03-07 (Actual); Primary Completion 2017-06-06 (Actual); Study Completion 2017-06-06 (Actual)

PRIMARY OUTCOMES:
Weight | 8 weeks
  Weight of subject in Kgs
MUAC | 8 weeks
  Mid Upper Arm Circumference in cms
TSF | 8 weeks
  Tricep Skin Fold thickness in mms

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Kashif Shafique, PhD, Study Director — Dow University of Health Sciences
Locations (1):
- Dow University of Health Sciences, Karachi, Sindh, Pakistan

IPD SHARING:
Plan to Share IPD: Undecided
If chosen for inclusion in meta analysis, Individual Participant Data (IPD) on outcome variables may be shared